CLINICAL TRIAL: NCT07335419
Title: PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD, CROSSOVER STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE EFFECT OF ITRACONAZOLE ON PF-07248144 PHARMACOKINETICS
Brief Title: A Study to Learn if Itraconazole Changes How the Body Processes PF-07248144 (Study Medicine)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4551006
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants
Keywords: Itraconazole; PF-07248144; Drug-Drug Interaction (DDI)
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-07248144 with and without Itraconazole (Experimental): Period 1; PF-07248144 single dose, oral tablet on Day 1. Period 2; Itraconazole oral solution once daily on Days 1-12 plus PF-07248144 single dose, oral tablet on Day 4.
  Period 1 and Period 2 will be separated with a washout of at least 14 days
  Interventions: Drug: PF-07248144; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-07248144 — Participants will receive PF-07248144 as a single dose, oral tablet on Day 1 of Period 1 and Day 4 of Period 2 with a washout period between two doses
Drug: Itraconazole — Participants will receive Itraconazole oral solution once daily on Days 1-12 in Period 2

SUMMARY:
The purpose of the study is to learn how itraconazole changes how the body processes the study medicine called PF-07248144. The study will also look at the safety, tolerability, and how PF-07248144 is changed and removed from the body after taking PF-07248144 alone compared to when it is taken with itraconazole.

Itraconazole can change how your body processes some medications so it may change the body's processing of PF-07248144. Multiple blood samples will be collected after each dose of PF-07248144 to determine how much PF-07248144 is in the blood at different times. This will help characterize the pharmacokinetics (pharmacokinetics helps us understand how the drug is changed and eliminated from your body after you take it) of PF-07248144 alone and when taken with itraconazole.

ELIGIBILITY:
Inclusion

* Female of nonchildbearing potential or males with 18 years of age or older, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead electrocardiograms
* Body mass index 18-32 kg/m2
* Total body weight >50 kg (110 lb)

Exclusion

* Pregnant female participants; breastfeeding female participants; female participants of childbearing potential; fertile male participants who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 103 days after the last dose of study intervention
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention
* Any prior use of epigenetic modifying agents
* Current use or anticipated need for food or drugs that are known moderate or strong inducers or inhibitors of CYP2C9 or CYP3A4, including their administration within 14 days or 5 half-lives of the strong inducers or inhibitors of CYP2C9 or CYP3A4, whichever is longer, prior to first dose of study intervention, during the treatment period, and within 10 days after the last dose of PF-07248144

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to extrapolated infinite time (AUCinf) for PF-07248144 | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours post-dose
Area under the concentration-time curve from time zero to time of last measurable concentration (AUClast) for PF-07248144 | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours post-dose
  AUClast will be used as the primary endpoint if AUCinf cannot be reliably estimated
Maximum observed plasma concentration (Cmax) for PF-07248144 | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours post-dose

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | From baseline up to 28 to 35 days post last study intervention dose
Number of participants with laboratory test abnormalities | From baseline up to 28 to 35 days post last study intervention dose
Number of participants with vital signs values meeting categorical summarization criteria | From baseline up to 28 to 35 days post last study intervention dose
Number of participants with clinically significant physical examination abnormalities | From baseline up to 28 to 35 days post last study intervention dose
Number of participants with treatment emergent clinically significant abnormal electrocardiogram (ECG) measurements | From baseline up to 28 to 35 days post last study intervention dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4551006